CLINICAL TRIAL: NCT06069622
Title: The Role of Glucagon-like Peptide 1 (GLP-1) Receptor Agonist Treatment of Overweight/Obese Individuals for Improving Adverse Cardiometabolic Phenotype Associated With CAV-1 Deficiency
Brief Title: Role of Caveolin 1 (CAV-1) Deficiency in Response to Glucagon-like Peptide 1 (GLP-1) Receptor Agonist Treatment
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Charles A. King Trust Postdoctoral Fellowship Program (Unknown)
Responsible Party: Principal Investigator, Ezgi Caliskan Guzelce, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2023P002452
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity
Keywords: GLP-1 receptor agonist; Weight loss; CAV-1; Blood pressure; ALDO
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Overweight and Obese individuals: A group of overweight and obese men and women whose body mass index (BMI) is ≥30.0 kg/m2 or ≥27.0 kg/m2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, prediabetes, dyslipidemia, obstructive sleep apnea whose treating clinicians have elected to start on semaglutide.
  Interventions: Diagnostic Test: 24-hour ambulatory blood pressure; Dietary Supplement: Liberal salt diet

INTERVENTIONS:
Diagnostic Test: 24-hour ambulatory blood pressure — 24-hour ambulatory blood pressure, blood, and urine will be obtained prior to semaglutide therapy and after 20 weeks of semaglutide therapy.
  Other Names: Blood collection; Urine collection
Dietary Supplement: Liberal salt diet — Participants will be on a liberal salt (about 200 mEq sodium/day) diet for 7 days.

SUMMARY:
Obesity has become an important public health issue that leads to insulin resistance, diabetes, hypertension, dyslipidemia, and cardiovascular diseases. Although weight loss with calorie restriction and increased physical activity improve these complications, many people fail these lifestyle interventions. Therefore, pharmacologic agents have been used for weight management in addition to lifestyle interventions. In the past few years, one of the widely used pharmacologic agents for weight management is Glucagon-like peptide 1 receptor agonists (GLP1 RAs). Overall, this class of medications improves both metabolic and cardiovascular profiles while causing weight loss, but their effects can vary between individuals. Therefore, it is essential to understand who will respond best to this therapy. Based on previous research on the interaction between a cell membrane molecule, caveolin-1, and glucagon-like peptide 1 receptor, we hypothesize that genetic variations in the caveolin-1 gene explain the variable cardiometabolic responses.

DETAILED DESCRIPTION:
Obesity is a chronic, multifactorial, and relapsing disease with an increasing prevalence that leads to insulin resistance, diabetes mellitus, hypertension, dyslipidemia, and cardiovascular diseases. Weight loss is known to improve metabolic and cardiovascular risk profiles. Although calorie restriction and increased physical activity represent the cornerstone of weight management treatment, clinical guidelines suggest adjunctive pharmacotherapy, particularly for adults with a BMI of 30 kg/m2 or greater or 27 kg/m2 or greater with coexisting conditions. Glucagon-like peptide 1 receptor agonists (GLP1 RAs) are highly effective in inducing weight loss in overweight and obese adults and have also been shown to improve cardiovascular outcomes. Elevated blood pressure (BP) is a well-known cardiovascular risk factor. Although GLP1 RAs improve insulin resistance, dyslipidemia, and type 2 diabetes, the beneficial effects of GLP1 RAs on BP are variable. This proposal's fundamental goal is to understand the mechanisms underlying this variable BP response to GLP1 RAs and investigate whether there is a variable response to weight loss.

Caveolin 1 is a protein on cell membrane that interacts with the GLP1 receptor and regulates its action. Our research laboratory previously demonstrated that a common polymorphism of the caveolin 1 (CAV1) gene (minor allele [C] at rs926198), which is associated with caveolin 1 deficiency, is strongly associated with higher BP and other components of the metabolic syndrome. This proposal will test the hypothesis that CAV-1 genotype will affect the CV and metabolic responses to treatment of overweight/obese individuals with a GLP-1 RA. Overall, demonstrating that a common variant in the CAV1 gene identifies the blood pressure and weight loss responses to GLP-1 RAs would be a very significant clinical outcome as GLP1 RAs use is rapidly increasing and would help lead to personalized therapy for obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, body mass index (BMI) ≥30.0 kg/m2 or ≥27.0 kg/m2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, prediabetes, dyslipidemia, obstructive sleep apnea,
* Normal screening laboratory values,
* Systolic BP < 160 mmHg and diastolic BP < 95 mmHg as determined from measurement during screening, using a random-zero device in the clinic and normal electrocardiogram, use of anti-hypertensive medications will be allowed except for mineralocorticoid receptor antagonists.

Exclusion Criteria:

* Diabetes mellitus,
* Treatment with a glucose-lowering agent(s) or anti-obesity medication within 90 days of screening,
* Treatment with a GLP-1 receptor agonist within 180 days,
* Current treatment with beta-blocker, or steroids,
* Pregnancy,
* Personal history of pancreatitis,
* Personal history of cholelithiasis,
* Previous surgical obesity treatment,
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma,
* Medical illness other than hypertension, prediabetes, obstructive sleep apnea, or dyslipidemia,
* Alcohol intake >12 oz. per week,
* Tobacco, or recreational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥18 years, men and women who have body mass index (BMI) ≥30.0 kg/m2 or ≥27.0 kg/m2 with the presence of at least one of the weight-related comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure response to GLP-1 RA treatment | 20 weeks
  The primary outcome will be the change (pre- treatment minus post-treatment) in mean 24-hour ambulatory systolic BP on a controlled dietary sodium intake in both CAV1 non-risk and risk genotypes.
Weight loss response to GLP-1 RA treatment | 20 weeks
  The primary outcome will be the mean percent change (pre- treatment minus post-treatment) in body weight in both CAV1 non-risk and risk genotypes.

SECONDARY OUTCOMES:
Aldosterone response to GLP-1 RA treatment | 20 weeks
  The secondary outcome will be changes in 24-hour urinary aldosterone levels in response to GLP-1 RA treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No